CLINICAL TRIAL: NCT02472483
Title: Effectiveness of TCC Followed by MBCT and Predictive Factors (Genetic, Clinical and Cognitive) Response
Acronym: TCC-MBCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult for recruting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D470
Record Dates: First submitted 2015-02-27; First posted 2015-06-16 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Bipolar Disorder; Anxious Disorder; Alcohol Dependence
MeSH Terms: conditions — Bipolar Disorder; Alcoholism | interventions — Cognitive Behavioral Therapy; Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- bipolar disorder (Experimental): Cognitive and Behavior Therapy (CBT) : 20-weeks CBT
  + Mindfulness Based Cognitive Therapy (MBCT) : 8-weeks MBCT
  Interventions: Behavioral: Cognitive and Behavior Therapy (CBT); Behavioral: Mindfulness Based Cognitive Therapy (MBCT)
- anxious disorders (Experimental): Cognitive and Behavior Therapy (CBT) : 20-weeks CBT
  + Mindfulness Based Cognitive Therapy (MBCT) : 8-weeks MBCT
  Interventions: Behavioral: Cognitive and Behavior Therapy (CBT); Behavioral: Mindfulness Based Cognitive Therapy (MBCT)
- alcohol disorder (Experimental): Cognitive and Behavior Therapy (CBT) : 20-weeks CBT
  + Mindfulness Based Cognitive Therapy (MBCT) : 8-weeks MBCT
  Interventions: Behavioral: Cognitive and Behavior Therapy (CBT); Behavioral: Mindfulness Based Cognitive Therapy (MBCT)

INTERVENTIONS:
Behavioral: Cognitive and Behavior Therapy (CBT) — 20-weeks CBT
Behavioral: Mindfulness Based Cognitive Therapy (MBCT) — 8-weeks MBCT

SUMMARY:
The purpose of this study is to determine whether a Cognitive and Behavioral group Therapy (CBT) + Mindfulness Based Cognitive Therapy (MBCT) decreased relapses and hospitalizations and improved outcomes (depressive and manic symptoms, self-esteem, and quality of life) in a large sample of refractory bipolar I patients on mood stabilizers.

DETAILED DESCRIPTION:
In recent years, various controlled studies showed that psychoeducational interventions have been effective in decreasing relapse and improving outcomes for bipolar disorders. However, samples were often small, compromising statistical power, and with a large variety of patients. The investigators therefore tested if a CBT group psychoeducation program + MBCT decreased relapses and improved outcomes in a large sample of refractory bipolar I patients on mood stabilizers. Patients were tested at recruitment, at 6-month follow-up CBT and at 2-month follow-up MBCT using clinical interviews and self-report questionnaires. The primary outcome measure of efficacy was relapse during the follow-up requiring either hospitalization, modification of treatment or HDRS ≥ 16 or MRS ≥ 6. The secondary outcome measure was symptomatic and functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Men and women
* Addressed to the CBT unit of the Clinique des Maladies Mentales et de l'Encéphale - CMME- (Sainte Anne Hospital)
* Having a bipolar I or II disorder (224 patients) or eating disorder (224 patients) : bulimia or discorder of use alcohol or gambling (224 patients)
* mood stabilizer treatment for more than six months, for bipolar patients
* Understanding and speaking French fluently
* Patient agreeing to participate and signing the consent form

Exclusion Criteria:

* Age <18 or> 65
* current manic, hypomanic, or depressive episode for bipolar patients
* Score on the Hamilton Depression Rating Scale - HDRS greater than or equal to 16
* Score on the Mania Rating Scale - MRS higher or equal to 6 for bipolar patients
* Schizophrenic disorder
* Severe somatic pathology (cancer, heart, kidney or respiratory failure, central neurological disorder), scalable, or are likely to be life-threatening in a period of less than one year
* Refusal of a mood stabilizer treatment for bipolar patients
* Inability to respond to assessment (eg failure or deterioration of mental ability.)
* No affiliation to a social security scheme
* Private topics of liberty by judicial or administrative decision
* Pregnant women

For bipolar patients, the presence of rapid cycling, family history of bipolar disorder, comorbid Axis I and II disorders, protective measures (curatorship or guardianship) are not exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2012-09-13 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Number of relapses (for bipolar disorders) | 22-months
  Number of relapses during 22-month

SECONDARY OUTCOMES:
Number of hospitalizations (for bipolar disorders) | 22-months
  Number of hospitalizations during 22-months
Number of days in an episode (for bipolar disorders) | 22-months
  Number of days in an episode during 22-months
Anxious symptomatology | 22-month
  Improvement of manic, depressive and/or anxious symptomatology during 22-month (scores MRS, HDRS, BDI,HARS, STAI)
Maniac symptomatology | 22-month
  Improvement of maniac, depressive and/or anxious symptomatology during 22-month (scores MRS, HDRS, BDI,HARS, STAI)
Depressive symptomatology | 22-month
  Improvement of maniac, depressive and/or anxious symptomatology during 22-month (scores MRS, HDRS, BDI,HARS, STAI)
Genetic polymorphisms | D0 (Inclusion)

CONTACTS AND LOCATIONS:
Overall Officials: Philip GORWOOD, MD., PhD, Principal Investigator — Centre Hospitalier Sainte-Anne
Locations (1):
- Centre Hospitalier Sainte Anne, Paris, France